CLINICAL TRIAL: NCT04226079
Title: Analysis of Volatile Organic Compound (VOC) in Exhaled Breath for the Detection of Gastrointestinal Bleeding
Brief Title: Volatile Organic Compounds (VOCs) of Exhaled Breath in Patients With GI Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunsoo Chung, Professor, Seoul National University Hospital
Other Study IDs: 1911-086-107
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Hemorrhage; Volatile Organic Compounds
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal control: Normal population with low prevalence of gastrointestinal bleeding who underwent EGD and CFS which revealed no abnormal finding.
  Interventions: Diagnostic Test: Collection of exhaled breath
- Patients with GI bleeding: Patients who visited emergency room and were highly suspected to have recent or active upper GI bleeding and scheduled for upper GI endoscopy.
  Interventions: Diagnostic Test: Collection of exhaled breath

INTERVENTIONS:
Diagnostic Test: Collection of exhaled breath — Collection of exhaled breath will be analyzed for specific volatile organic compounds which show different distribution between groups

SUMMARY:
Cross sectional case-control study investigating the difference of volatile organic compound in the exhaled breath of the patients with GI bleeding and normal population.

DETAILED DESCRIPTION:
This study investigates the difference of volatile organic compound in the exhaled breath of the patients with GI bleeding and normal population. We aimed to find out the biomarkers for GI bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 20 and 80
* Low possibility of gastrointestinal bleeding was proven by esophagogastroduodenoscopy and colonoscopy which were performed within 1 year.
* NSAID non-user (within 1 months before the date of inclusion)

Exclusion Criteria:

* Diagnosis of malignancy diagnosed within 5 years
* Past medical history of chronic liver disease, chronic kidney disease, chronic lung disease, chronic bronchial disease, asthma
* Surgical history of any kind of gastrectomy
* Surgical history of any kind of lung resection which could impact the patient's lung function.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Adults aged 20-80
  * Patients who visited emergency room and suspected to have recent or active gastrointestinal bleeding
  * Patients who are scheduled to undergo esophagogastroduodenoscopy.
  Exclusion Criteria:
  * Diagnosis of malignancy diagnosed within 5 years
  * Past medical history of chronic liver disease, chronic kidney disease, chronic lung disease, chronic bronchial disease, asthma
  * Surgical history of any kind of gastrectomy
  * Surgical history of any kind of lung resection which could impact the patient's lung function.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
VOC Patterns | 1 day of 1st emergency room (ER) visit for GI bleeding
  Patterns of volatile organic compounds recognized by sensor array

SECONDARY OUTCOMES:
Measurement of VOC | 1 day of 1st emergency room (ER) visit for GI bleeding
  Qualitative and quantitative assay of volatile organic compounds by GC-MS
Change of VOC patterns | 2nd visit (about 2weeks apart from 1st visit)
  Change of the patterns of volatile organic compounds recognized by sensor array after recovery from GI bleeding

CONTACTS AND LOCATIONS:
Overall Officials: HYUNSOO CHUNG, M.D., Study Chair — Seoul National University Hospital
Locations (1):
- Jin Ju Choi, Seoul, Gyunggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided